CLINICAL TRIAL: NCT01464320
Title: A Phase 1b, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of a Single-Dose of ABT-614 and the Effect of ABT-614 on Glomerular Filtration Rate in Subjects With Type 2 Diabetes and Chronic Kidney Disease With Albuminuria
Brief Title: A Study to Evaluate the Safety and Tolerability of ABT-614 and Its Effect on Kidney Function in Subjects With Type 2 Diabetes and Chronic Kidney Disease With Protein in Their Urine.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: M13-107
Record Dates: First submitted 2011-11-01; First posted 2011-11-03 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-04

CONDITIONS: Type 2 Diabetics, Chronic Kidney Disease, Protein in Urine
Keywords: Safety; Type 2 diabetes; Kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Proteinuria; Diabetes Mellitus, Type 2; Kidney Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ABT-614 (Experimental)
  Interventions: Drug: ABT-614
- Placebo Comparator (Placebo Comparator)
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: ABT-614 — Active
  Arms: ABT-614
Drug: Placebo Comparator — Placebo
  Arms: Placebo Comparator

SUMMARY:
To assess the safety, tolerability and pharmacokinetics of ABT-614 in subjects with type 2 diabetes and chronic kidney disease with albuminuria and to determine whether ABT-614 reduces glomerular filtration rate.

DETAILED DESCRIPTION:
This Phase 1b, single-site, double-blind, randomized, placebo-controlled study will be conducted in three Periods; Baseline, Dosing and Outpatient. Eligible adult male and female subjects with type 2 diabetes and CKD (chronic kidney disease) with albuminuria will be selected to participate.

Eighteen subjects will be selected to participate in the Baseline Period to ensure that 16 subjects are enrolled in the Dosing Period. Subjects who are eligible from Screening will be confined to the study site beginning on Day -2 (the day before the Baseline Period infusion). On Day -1, subjects will be administered an iothalamate infusion to measure baseline GFR (glomerular filtration rate). Subjects who continue to be eligible on Day 1 will be randomized in a 1:1 ratio to receive either a 10 mg dose of ABT-614 or matching placebo daily, for 15 days.

On Day 15 subjects will be administered a second iothalamate infusion. Plasma and urine samples for ABT-614 and iothalamate will be collected. Subjects will be released from confinement on Day 20 after the completion of all study procedures including the 120-hour blood sample collection. Thereafter, subjects will return for outpatient visits on Days 25 and 30 as well as 30 days after the last dose of study drug. A ± 2 day window will be permitted on the 30-day Follow-up Visit to accommodate subject scheduling.

ELIGIBILITY:
Inclusion Criteria

1. Male or female aged between 19 and 70 years, inclusive, at time of consent.
2. Type 2 diabetes receiving at least one anti-diabetic medication for at least one year at the time of Screening.
3. Hemoglobin A1c < 12% at the time of Screening.
4. Estimated glomerular filtration rate ≥ 30 mL/min calculated by the Cockcroft-Gault Formula at the time of Screening.
5. Urinary albumin to creatinine ratio 100 to 5000 mg/g creatinine at the time of Screening.

Exclusion Criteria

1. History of unusual or allergic reaction to iodine, to products containing iodine (for example., iodine containing foods) or to other radio-opaque agents.
2. Subject history of epileptic seizures or convulsions.
3. Clinically significant cardiac disease or family history of long-QT syndrome and/or subject and/or family history of unexplained, sudden cardiac death. History of myocardial infarction or coronary artery bypass graft is not exclusionary if occurrence is ≥ 12 months prior to the administration of study drug and the subject does not have conduction abnormality and has been stable without intervention, symptoms of ischemia or an increase in cardiovascular medications. Electrocardiography (ECG) should be compared with historical to ensure no new clinically significant changes have occurred.
4. History of gastric surgery, cholecystectomy, vagotomy, bowel resection or any surgical procedure that might interfere with gastrointestinal motility, potential hydrogen (pH) or absorption.
5. Clinically significant respiratory (except mild asthma), gastrointestinal, hematologic, neurologic, thyroid or any uncontrolled medical illness or psychiatric disease or disorder.
6. Screening ECG with clinically significant abnormalities and/or confirmed Screening QTcF prolongation more than 430 milliseconds for males and 450 milliseconds for females or ECG with second or third degree atrioventricular block.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Change in drug concentration | Day -1 (Baseline) and up to Day 15
  Blood and urine tests
Change in glomerular filtration rate | Day -1 (Baseline) and up to Day 15
  Blood and urine tests

SECONDARY OUTCOMES:
Change in urinary albumin excretion | Day -1 (Baseline) and up to Day 15
  Urine tests

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Andress, MD, Study Director — Renal Global Project Team, Abbott Laboratories
Locations (1):
- Site Reference ID/Investigator# 63442, Miami, Florida, United States